CLINICAL TRIAL: NCT02648984
Title: Ad Hoc Analysis for the Evaluation of Dynamic Pulmonary Vascular Resistance in Patients With a Closed Ventricular Septal Defect
Brief Title: Evaluation of Dynamic Pulmonary Vascular Resistance in Patients With Closed Ventricular Septal Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Werner Budts, Werner Budts, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S56272
Record Dates: First submitted 2015-12-30; First posted 2016-01-07 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Vascular Disease
Keywords: Pulmonary vascular disease

ARMS (2):
- Patient group (Other): Patients with ventricular septal defect
  Interventions: Other: The intervention is performing an exercise test
- Control group (Other): Healthy control subjects
  Interventions: Other: The intervention is performing an exercise test

INTERVENTIONS:
Other: The intervention is performing an exercise test — Patients and controls will undergo a bicycle stress echocardiography and a cardiopulmonary exercise test

SUMMARY:
Pulmonary arterial hypertension (PAH) in patients with congenital heart disease usually develops secondary to chronic volume overload of the pulmonary circulation following left to right shunt. This overload leads to elevated pulmonary artery pressure (PAP) and later to increased pulmonary vascular resistance (PVR), leading to right ventricular dysfunction, considerable morbidity and even mortality.

Since PAH nowadays is mostly detected when symptoms occur and PAP are elevated, the disease already evolved to an advanced stage and treatment is often initiated too late. Our research group standardized the technique for the detection of early pulmonary vascular disease by bicycle stress echocardiography. The investigators now aim to assess this exercise technique in a group of patients with ventricular septal defect.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) in patients with congenital heart disease usually develops secondary to chronic volume overload of the pulmonary circulation following left to right shunt. This overload leads to elevated pulmonary artery pressure (PAP) and later to increased pulmonary vascular resistance (PVR). PAH may lead to right ventricular and right atrial dysfunction, which may implicate considerable morbidity and even mortality.

Since PAH nowadays is mostly detected when symptoms occur and PAP are elevated, the disease already evolved to an advanced stage and treatment is often initiated too late. Our research group standardized the technique for the detection of early pulmonary vascular disease by bicycle stress echocardiography. Exercise-induced pulmonary hypertension has been recognised as a clinical entity, but is not included in the current guidelines on pulmonary hypertension. Further research in this area might imply the need for revision of the current PAH detection and treatment strategy.

By performing stress echocardiography and cardiopulmonary exercise testing, the investigators want to reach the following objectives:

* To answer the question whether the abnormal increase in PAP during exercise, seen in patients with late atrial septal defect (ASD) type secundum closure, is also present in congenital heart disease (CHD) patients who were treated for other shunt lesions.
* To apply this early detection technique in a broader population of CHD patients and to better define the predictive value of an elevated PVR during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with ventricular septal defect (VSD) repair at least 6 months before study enrolment
* No discrimination in type of VSD repair will be made (percutaneous or surgical)
* Subjects must be able to perform exercise testing

Exclusion Criteria:

* Other congenital heart disease
* PAH of any aetiology other than VSD
* Inclusion in other treatment protocols
* Impairment of organic function (renal, hepatic)
* Arterial hypotension (systolic blood pressure < 85 mmHg)
* Anaemia (Hb < 10 g/dl)
* Thrombocytopenia (< 50000/µl)
* Significant valvular disease, other than tricuspid or pulmonary regurgitation
* Chronic lung disease or total lung capacity < 80% of predicted value
* History of pulmonary embolism
* Cyanotic patients, patients in an unstable condition and patients who have to undergo re-intervention during the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery pressure - flow plot | Through study completion, an average of 1,5 years for the first testing, an additional 1 year for the retesting

SECONDARY OUTCOMES:
Maximal Oxygen Uptake | Through study completion, an average of 1,5 years for the first testing, an additional 1 year for the retesting

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium